CLINICAL TRIAL: NCT06365684
Title: Sodium Zirconium Cyclosilicate to Allow Liberal Fruit and Vegetable Intake for Patients With CKD Stage 3b and 4
Acronym: LIBRAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, JorisRotmans, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 133548; 2023-507823-52 (EudraCT Number)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-04

CONDITIONS: Hyperkalemia; Diet Modification; Chronic Kidney Disease; Sodium Zirconium Cyclosilicate
Keywords: Fruit, vegetables and nuts; increase dietary potassium intake; Lokelma; Sodium zirconium Cyclosilicate; Chronic Kidney disease; Safety
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: Single center, cross-over randomized clinical trial with non-inferiority design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potassium enriched diet (Experimental): Patients with chronic kidney disease stage 3b to 4 will be treated for 6 weeks with a potassium enriched diet (adding +40mmol/day in the form of fruits/vegetables/nuts)
  Interventions: Drug: Sodium zirconium cyclosilicate
- Regular diet (No Intervention): Patients with chronic kidney disease stage 3b to 4 will followed for 6 weeks, during their regular diet

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — In the case of hyperkalemia patients will be treated with Sodium zirconium cyclosilicate to allow the continuation of potassium enriched diet. In case hyperkalemia arises in the control group, patients will be treated with Sodium zirconium cyclosilicate as well.
  Other Names: Lokelma
  Arms: Potassium enriched diet

SUMMARY:
Rationale: Several studies have shown that higher urinary potassium excretion (as proxy for potassium intake) is associated with better kidney outcomes, lower blood pressure and improved survival. These associations are also observed in patients with (advanced) CKD. However, application in daily practice in patients with CKD, is impaired by the risk of hyperkalemia, due to metabolic acidosis and impaired renal potassium excretion in these patients. As a consequence, patients with CKD are advised to restrict their intake of fruit and vegetables, as these healthy food components are important sources of dietary potassium. This is particularly undesirable for patients with CKD in view of the very high risk of cardiovascular disease.

Concomitant use of sodium zirconium cyclosilicate (SZC) could allow a more liberal intake of fruit and vegetables for patients with CKD, as SZC effectively treats hyperkalemia and counteracts metabolic acidosis [1]. With this strategy, the beneficial effects of potassium in fruits and vegetables on (vascular) health could also become accessible to patients with CKD.

Objective: To demonstrate that a potassium-rich diet, including the use of SZC as potential rescue treatment (in case of hyperkalemia), does not result in an unacceptable rise in plasma potassium (i.e. max rise of 0.5 mmol/L and no hyperkalemia). Study Design: Investigator initiated, single center, cross-over randomized clinical trial with non-inferiority design (14 weeks, 2 groups: regular diets vs. diet with potassium rich fruits and vegetables with sodium zirconium cyclosilicate if necessary) Study population: Outpatients ( age ≥ 18 years ) with chronic kidney disease stage IIIb/IV and use of inhibitor of the renin-angiotensin system (RASi).

Intervention: Addition of fruit- and vegetables that contain 40 mmol of potassium on top of regular diet. Addition of SZC after 1 week in case hyperkaliemia develops (serum potassium > 5,5 mmol/L). Weekly measurement of plasma potassium and dose adjustment of SZC if needed

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney disease, stage 3 to 4b (eGFR 44-15 ml/min/1.73m^2)
* Use of inhibitor of the renin-angiotensin system

Exclusion Criteria:

* Hyperkaliemia (plasma potassium > 5.5 mmol/L) at baseline or at the start of potassium enriched diet
* Use of potassium binders at baseline or at the start of potassium enriched diet
* Use of dual RAAS-blockade, mineralocorticoid receptor blockers or potassium-sparing diuretics
* Use of calcineurin inhibitors
* Use of trimethoprim and sulfamethoxazole
* Patients with a previous history of ventricular cardiac arrhythmia
* Patients with a prolonged QTc time on ECG
* Kidney transplantation patients
* Patients with a life expectancy of < 6 months
* Incapacitated subjects or subjects who are deemed unfit to adequately adhere to instructions from the research team
* Women who are pregnant, breastfeeding or considering pregnancy in the coming 6 months.
* Hypersensitivity to SCZ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The difference of serum potassium at baseline and after six weeks of treatment with potassium enriched diet (non-inferiority design) compared to the control group. With an intention to treat analysis. | 6 weeks

SECONDARY OUTCOMES:
Ambulatory blood pressure (average systolic and diastolic blood pressure over 24 hours) | 6 weeks
24 hours albuminuria | 6 weeks
urinary potassium (mmol/l) | 6 weeks
Plasma bicarbonate | 6 weeks
Quality of life, using SF36 questionnaire | 6 weeks
  36-Item Short Form Survey. Scoring can range from 0 to 100. Higher scores indicate better health status
Effect on stool (assessed with Bristol Stool Chart) | 6 weeks
  Scoring can range form 1 to 7. Where score of 1 indicates obstipation, score of 4 indicates normal defecation and 7 indicates watery defecation.
Difference in serum potassium one week after start of study (SCZ free period) | 6 weeks
Per protocol analysis of difference in serum potassium after six week (end of study) | 6 weeks
Incidence of severe hyperkalemia (serum potassium above 6.5 mmol/l or above 6.0 with ECG features of hyperkalemia) | 6 weeks
Incidence of hyperkalemia (serum potassium above 5.5 mmol/l) | 6 weeks
Necessity for treatment of hyperkalemia | 6 weeks
urinary sodium (mmol/l) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided